CLINICAL TRIAL: NCT02518711
Title: A Randomized Controlled Trial Into the Effectiveness of a Behavioral Teacher Program Targeting ADHD Symptoms
Brief Title: Effectiveness Study of a Behavioral Teacher Program Targeting ADHD Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: Stichting Kinderpostzegels Nederland (Unknown); Nederlandse Stichting voor het Gehandicapte Kind, The Netherlands (Unknown); Stichting Weeshuis der Doopsgezinden, The Netherlands (Unknown); Stichting Zonnige Jeugd, The Netherlands (Unknown)
Responsible Party: Principal Investigator, Betty Veenman, MSc, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METc VUmc 2011/196; 5930790 (Other Grant/Funding Number: KPZ); 20110028 (Other Grant/Funding Number: NSGK)
Record Dates: First submitted 2015-08-05; First posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: symptoms of ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral teacher program (Experimental): The behavioral teacher program was used by the participant's teacher in the classroom during 18 weeks.
  Interventions: Behavioral: Behavioral Teacher Program
- Control group (No Intervention): Children within the control group did not receive the behavioral teacher program but were allowed to receive regular care

INTERVENTIONS:
Behavioral: Behavioral Teacher Program — This program was based on the evidence-based Summer Treatment Program (MTA Cooperative Group, 1999), involving psycho-education for the teacher and universal and individual behavioral techniques that focused on classroom structure and contingency management
  Arms: Behavioral teacher program

SUMMARY:
The goal of this study was to investigate the effectiveness of a behavioral teacher program addressing symptoms of Attention-Deficit Hyperactivity Disorder (ADHD) in the classroom.

DETAILED DESCRIPTION:
Background:

Most behavioral teacher programs involve intensive and expensive teacher trainings by health care specialists, which may limit successful large-scale implementation. This behavioral program, on the contrary, involves a self-containing manual that does not require expert training in order to increase the likelihood of successful implementation (if proven effective). The aim was to investigate the program's effects on behavioral, socio-emotional and school functioning in primary school children.

Methods:

Children with ADHD symptoms were randomly assigned at school level to the intervention condition (receiving the program during 18 weeks) or control group (not receiving the program but who were allowed to receive care as usual).

Measures to assess program's effectiveness:

* Strengths and Weaknesses of ADHD-symptoms and Normal Behavior,
* Strengths and Difficulties Questionnaire
* Social Skills Rating Scale
* Spence Children's Anxiety Scale
* Classroom Observation Code
* Actigraphy
* Sociometric measures (peer nomination and peer rating)
* Dutch arithmetic test (Tempo-Test-Rekenen)
* reading test (Drie-Minuten-Toets) and writing test (PI-dictee).

Additional measures:

* Wechsler Intelligence Scale for Children (Block Design and Vocabulary; used to estimate IQ);
* Sensitivity to Punishment and Sensitivity to Reward Questionnaire and several neuropsychological computer tasks

ELIGIBILITY:
Inclusion Criteria:

* sub-threshold or clinical level of ADHD symptoms as observed by participant's teacher through the Dutch version of the Disruptive Behavior Disorders Rating Scale (Pelham, Gnagy, Greenslade, & Milich, 1992)
* at least one clinical and three sub-threshold ADHD symptoms as measured by the Teacher Telephone Interview (Holmes et al., 2004), a semi-structured interview which is based on the Diagnostic and Statistical Manual of Mental Disorders (American Psychiatric Association, 2000)

Exclusion Criteria:

* (medication) treatment for ADHD at study entry or in preceding 6 months;
* neurological or severe physical condition
* IQ < 80 based on a short version of the Wechsler Intelligence Scale for Children (Block Design and Vocabulary; Legerstee, van der Reijden-Lakeman, Lechner-van der Noort, & Ferdinand, 2004; Hrabok, Brooks, Fay-McClymont, & Sherman, 2014)
* participant enrolled in a daily contingency management program or other teacher program targeting behavior or social problems at study entry or in the preceding month
* Maximum of 2 children per classroom and 5 classrooms per school (in order to limit teachers' burden and increase heterogeneity of teacher and classroom settings)

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2011-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Strengths and Weaknesses of ADHD-symptoms and Normal Behavior Scale (SWAN; Young, Levi, Martin, & Hay, 2009) | 6 weeks and 18 weeks after baseline assessment
  The teacher and parent version of the SWAN were used
Change from Baseline in Strengths and Difficulties Questionnaire (SDQ; Van Widenfelt, Goedhart, Treffers, & Goodman, 2003) | 6 weeks and 18 weeks after baseline assessment
  The teacher and parent-version of the SDQ were administered, using the following subscales: ADHD, Conduct Problems, Internalizing Behavior (combining Emotional Symptoms and Peer Problems), and Impact On Daily Functioning
Change from Baseline in hyperactivity during school hours using Actigraphy (Cambridge Neurotechnology, 2008) | 6 weeks and 18 weeks after baseline assessment
  It concerned an actigraph worn on the wrist of the non-dominated hand during 5 school days
Change from Baseline in Disruptive Classroom Behavior measured by the Classroom Observation Code (COC; Abikoff, Gittelman, & Klein, 1980) | 6 weeks and 18 weeks after baseline assessment
  The observation was performed by well-trained psychology students not involved in treatment delivery. Each participant was observed twice on the same school day for 8 minutes, using the average score as outcome measure

SECONDARY OUTCOMES:
Change from Baseline in Social Skills Scale of the Social Skills Rating Scale (SSRS; Merrell & Popinga, 1994) | 6 weeks and 18 weeks after baseline assessment
  The teacher and parent version of the SSRS were used
Change from Baseline in Spence Children's Anxiety Scale (SCAS) | 6 weeks and 18 weeks after baseline assessment
  SCAS is a self-report administered to the child
Change from Baseline in Sociometric Measure (Bukowski, Cillessen, & Velasquez, 2012) | 6 weeks and 18 weeks after baseline assessment
  The sociometric measure includes both a peer nomination and a peer rating scale
Change from Baseline in Performance on Dutch Reading Test (Drie-Minuten Toets; Verhoeven, 1995) | 6 weeks and 18 weeks after baseline assessment
Change from Baseline in Performance on Dutch Writing Test (PI-dictee; Geelhoed & Reitsma, 2000) | 6 weeks and 18 weeks after baseline assessment
Change from Baseline in Performance on Dutch Arithmetic Test (Tempo-Test Rekenen; De Vos, 1992) | 6 weeks and 18 weeks after baseline assessment
Teacher's treatment fidelity averaged over 18 similar checklists (self-constructed), containing 13 items on a 3-point Likert scale regarding the use of each intervention element (0=not used or inadequate use, 1=adequate use, and 2=good use) | 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, and 18 weeks after start of the intervention
  Only teachers in the intervention group needed to fill in this rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Oosterlaan, PhD, Principal Investigator — VU University of Amsterdam

REFERENCES:
- [Background] Durlak JA, DuPre EP. Implementation matters: a review of research on the influence of implementation on program outcomes and the factors affecting implementation. Am J Community Psychol. 2008 Jun;41(3-4):327-50. doi: 10.1007/s10464-008-9165-0. PMID 18322790
- [Background] Han SS, Weiss B. Sustainability of teacher implementation of school-based mental health programs. J Abnorm Child Psychol. 2005 Dec;33(6):665-79. doi: 10.1007/s10802-005-7646-2. PMID 16328743
- [Background] A 14-month randomized clinical trial of treatment strategies for attention-deficit/hyperactivity disorder. The MTA Cooperative Group. Multimodal Treatment Study of Children with ADHD. Arch Gen Psychiatry. 1999 Dec;56(12):1073-86. doi: 10.1001/archpsyc.56.12.1073. PMID 10591283
- [Background] Pelham WE Jr, Gnagy EM, Greenslade KE, Milich R. Teacher ratings of DSM-III-R symptoms for the disruptive behavior disorders. J Am Acad Child Adolesc Psychiatry. 1992 Mar;31(2):210-8. doi: 10.1097/00004583-199203000-00006. PMID 1564021
- [Background] Holmes J, Lawson D, Langley K, Fitzpatrick H, Trumper A, Pay H, Harrington R, Thapar A. The Child Attention-Deficit Hyperactivity Disorder Teacher Telephone Interview (CHATTI): reliability and validity. Br J Psychiatry. 2004 Jan;184:74-8. doi: 10.1192/bjp.184.1.74. PMID 14702231
- [Background] Legerstee JS, van der Reijden-Lakeman IA, Lechner-van der Noort MG, Ferdinand RF. Bruikbaarheid verkorte versie wisc-rn in de kinderpsychiatrie. Kind en adolescent. 2004;25(4):178-82. doi: 10.1007/BF03060926.
- [Background] Hrabok M, Brooks BL, Fay-McClymont TB, Sherman EM. Wechsler Intelligence Scale for Children-fourth edition (WISC-IV) short-form validity: a comparison study in pediatric epilepsy. Child Neuropsychol. 2014;20(1):49-59. doi: 10.1080/09297049.2012.741225. Epub 2012 Dec 10. PMID 23216421
- [Background] Young DJ, Levy F, Martin NC, Hay DA. Attention deficit hyperactivity disorder: a Rasch analysis of the SWAN Rating Scale. Child Psychiatry Hum Dev. 2009 Dec;40(4):543-59. doi: 10.1007/s10578-009-0143-z. Epub 2009 May 20. PMID 19455417
- [Background] Merrell KW, Popinga MR. The alliance of adaptive behavior and social competence: an examination of relationship between the scales of Independent Behavior and the Social Skills Rating System. Res Dev Disabil. 1994 Jan-Feb;15(1):39-47. doi: 10.1016/0891-4222(94)90037-x. PMID 8190971
- [Background] CambridgeNeurotechnology. The Actiwatch User Manual. Cambridge, 2008.
- [Background] Abikoff H, Gittelman R, Klein DF. Classroom observation code for hyperactive children: a replication of validity. J Consult Clin Psychol. 1980 Oct;48(5):555-65. doi: 10.1037//0022-006x.48.5.555. No abstract available. PMID 7410654
- [Background] Bukowski WM, Cillessen A, Velasquez A. Peer ratings. In: Laursen B, Little T, Card A, editors. Handbook of developmental research methods. New York: The Guilford Press; 2012. p. 211-28.
- [Background] De Vos T. Tempo-Test-Rekenen. Handleiding. [Tempo Test Arithmetic. Manual]. Nijmegen: Berkhout; 1992.
- [Background] Verhoeven L. Drie Minuten Toets Handleiding.[Three Minutes Test Manual]. Arnhem, The Netherlands: CITO. 1995.
- [Background] Geelhoed J, Reitsma P. PI-dictee. Handleiding. Lisse: PI Research Duivendrecht, Swets & Zeitlinger B.V.; 2000.
- [Derived] Veenman B, Luman M, Oosterlaan J. Moderators Influencing the Effectiveness of a Behavioral Teacher Program. Front Psychol. 2018 Mar 13;9:298. doi: 10.3389/fpsyg.2018.00298. eCollection 2018. PMID 29593604
- [Derived] Veenman B, Luman M, Oosterlaan J. Further Insight into the Effectiveness of a Behavioral Teacher Program Targeting ADHD Symptoms Using Actigraphy, Classroom Observations and Peer Ratings. Front Psychol. 2017 Jul 11;8:1157. doi: 10.3389/fpsyg.2017.01157. eCollection 2017. PMID 28744244